CLINICAL TRIAL: NCT04259658
Title: Phase II Investigation of the Histopathologic Effect of Calcium Electroporation on Cancer in the Skin (CAEP-B)
Brief Title: Histopathologic Effect of Calcium Electroporation on Cancer in the Skin
Acronym: CAEP-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-114-2019
Record Dates: First submitted 2020-01-21; First posted 2020-02-06 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: calcium; electroporation; tumor infiltrating lymphocytes; cancer; metastases
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective phase II clinical study: Patients with cutaneous metastases will be recruited at the Department of Oncology, Zealand University Hospital (ZUH). One cohort of 24 patients with respectively disseminated breast cancer or other solid tumour malignancies, will be included. This will be a non-randomized trial.
  All patients will have been offered the standard of care and all available alternatives before entering the protocol. Calcium electroporation will not be compared to other means of treatment.
  All patients will be treated once and patients with over 3 metastases will be offered retreatment of some of their metastases. A maximum of 2 treatments per patient will be conducted with an interval of minimum 4 weeks. The patients will be followed with regular examinations for 3 months, starting from first treatment day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcium electroporation treatment (Experimental): Experimental treatment with calcium electroporation for cutaneous metastases.
  Interventions: Combination Product: Calcium electroporation

INTERVENTIONS:
Combination Product: Calcium electroporation — Patients with cutaneous metastases will be treated with calcium electroporation.

SUMMARY:
In this phase II study we investigate the effect of calcium electroporation on cancer in the skin investigated by histopathology.

DETAILED DESCRIPTION:
In this non randomized phase II study, we will explore histopathological tumour cell death mechanisms in 24 patients with breast cancer metastases or other cutaneous or subcutaneous malignancy. The primary endpoint of the biopsy study is to evaluate differences in tumour infiltrating lymphocyte (TIL) population in tissue samples from treated cancer tumours two days after calcium electroporation treatment compared to samples taken on the day of treatment before the calcium electroporation procedure. TIL content in biopsies will be evaluated by pathological examination and specified in percent of cells. Patients will be followed up to 3 months and depending on number of treated tumors, biopsies will be taken at different timepoints after one or two treatments with calcium electroporation. Other analyses will include differences regarding tumour type, immune marker expression levels over time, vascular effects and regressive changes as well as examining changes in systemic immunological markers.

ELIGIBILITY:
Inclusion Criteria:

* Trial subject must be able to understand the participant information.
* Histologically verified cutaneous or subcutaneous, primary or secondary cancer of any histology.
* The patient can undergo any simultaneous medical treatment (endocrine therapy, chemotherapy, immunotherapy etc.).
* The patient can undergo radiation therapy during the study period, provided that the treatment field does not involve the treated area.
* Performance status ECOG/WHO ≤2
* At least one cutaneous or subcutaneous tumour measuring at least 5 mm.
* Both men and women who are sexually active must use safe contraception (contraceptive coil, deposit injection of gestagen, subdermal implantation, hormonal vaginal ring or transdermal patch.)
* Signed informed consent.

Exclusion Criteria:

* Pregnancy or lactation
* Allergy to local anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
The effect of calcium electroporation on tumor infiltrating lymphocyte (TIL) population. | 2 days
  The primary endpoint of this study is to evaluate differences in TIL population in tissue samples from treated cancer tumours two days after calcium electroporation treatment compared to before treatment (biopsy taken on the day of treatment before the calcium electroporation procedure). TIL content in biopsies will be evaluated by pathological examination and expressed as percent of cells.

SECONDARY OUTCOMES:
Changes in immune markers | 3 months
  Protein expression levels of immune markers e.g. markers for the innate and adaptive immune system and markers of the STING pathway compared from before treatment and at different timepoints up to 3 months.
Tumour inflammation signature (TIS) | 3 months
  Gene expression signatures including the 18-gene TIS will be calculated as a weighted linear average of the constituent genes.
Molecular subtype classification | 3 months
  Gene expression profiling according to tumour histology.
Size of lesion | 3 months
  To clinically measure changes in lesion size 1, 2 and 3 months after treatment using caliper measurement. Changes in size due to biopsies will be accounted for.
TIL population and tumour type | 3 months
  To describe any relation between change in TIL population (percentage of cells) and tumour type before and after calcium electroporation.
Tumour regression | 3 months
  To describe presence of regressive changes including necrosis at different timepoints (percentage of tissue).
Residual tumour | 3 months
  To describe presence of residual tumour (yes/no) and description of topographical location.
Vascular effects | 3 months
  To investigate vascular effects of calcium electroporation including changes in capillary structures by histochemical staining for endothelial biomarkers CD31 and/or CD34.
Clinical response to intervention | 3 months
  To document evolution of tumours before and after treatment using digital photography including a ruler.
Complete response at patient level | 3 months
  To sum number of patients with complete response after one or two treatments, respectively. Complete response will be defined as disappearance of all target lesions.
Complete disappearance of treated lesions (in relation to all lesions treated) | 3 months
  To sum number of lesions across all patients with complete remission after one or two treatments, respectively (expressed at percentage of all treated lesions).
Tumour type | 3 months
  To establish number of treated tumours with complete response depending on tumour type.
Systemic immunologic response | 3 months
  To detect signs of systemic immunologic response from any routine scans before and after treatment in the inclusion period.
Importance of previous irradiation | 3 months
  To investigate differences in effect depending whether the treated tumour was in a previously irradiated area.
Adjacent non-tumour tissue | 3 months
  To evaluate effect on adjacent non-tumour tissue.
PD-L1 expression over time | 3 months
  To assess PD-L1 expression over time by biopsy.
Relation between change in PD-L1 expression and response | 3 months
  To investigate any relation between change in PD-L1 expression and tumour response.
PD-L1 expression in relation to cell types | 3 months
  To describe PD-L1 expression in relation to cell types found in the tumour environment
PD-L1 expression of different tumour histologies | 3 months
  To describe PD-L1 expression on different cell types of the different tumour histologies investigated.
Western blotting | 3 months
  To examine frozen tissues samples by western blotting in order to support any of the above mentioned endpoints.
Systemic immune factors after calcium electroporation | 3 months
  Blood samples may be analyzed for NK cell- and T-cell gene expression levels. Levels before and after treatment will be compared.
Current measurement | 1 month
  To measure current during treatment as indicated by the pulse generator.
PCR | 3 months
  To examine frozen tissues samples by PCR. Relevant gene expression will be compared before and after treatment in breast cancer and non breast cancer samples.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Dept. of Clinical oncology and Palliative Care, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No